CLINICAL TRIAL: NCT04910789
Title: A Prospective, Multicenter, Randomized, Controlled Study Comparing Surgical Efficacy Between Transhiatal/Transabdominal and Thoracoabdominal Approach for Patients With Siewert II Adenocarcinoma of Esophagogastric Junction
Brief Title: Transhiatal/Transabdominal Approach Compare With Thoracoabdominal Approach for Siewert II Adenocarcinoma of Esophagogastric Junction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, Prof., Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2AEG
Record Dates: First submitted 2021-05-20; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Adenocarcinoma of Esophagogastric Junction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracoabdominal approach (Experimental): Radical surgery should be finished via Thoracoabdominal approach.
  Interventions: Procedure: thoracoabdominal approach
- Transhiatal/transabdominal approach (Active Comparator): Radical surgery should be finished via transhiatal/transabdominal approach.
  Interventions: Procedure: transhiatal/transabdominal approach

INTERVENTIONS:
Procedure: transhiatal/transabdominal approach — Radical surgery should be finished via transhiatal/transabdominal approach
  Arms: Transhiatal/transabdominal approach
Procedure: thoracoabdominal approach — Radical surgery should be finished via thoracoabdominal approach
  Arms: Thoracoabdominal approach

SUMMARY:
To compare transhiatal / transabdominal approach with thoracoabdominal approach for Siewert II adenocarcinoma of esophagogastric junction

DETAILED DESCRIPTION:
Objective: To compare the safety and clinical efficacy between transhiatal/transabdominal and thoracoabdominal approach for Siewert Ⅱ adenocarcinoma of esophagogastric junction.

Methods: A prospective, multi-center, randomized, controlled study will be performed. Patients who meet the eligibility criteria will be registered in the study and undergo radical surgery via transhiatal/transabdominal or thoracoabdominal approach. The data of preoperative, intraoperative, postoperative and follow-up will be recorded and analyzed.

The primary endpoints :3-year disease-free survival. The secondary endpoints:(1) Surgery and oncology indicators ;(2) The incidences of postoperative complications and mortality.

ELIGIBILITY:
Inclusion Criteria:

* 1.18~75 years old
* 2.The tumor center located at the esophagogastric junction(EGJ) line from 1cm above to 2cm below(SiewertⅡ) .
* 3.Histological diagnosis of adenocarcinoma
* 4. American Society of Anesthesiologists(ASA) physical status class is less than or equal to 3
* 5.Informed consent of patients

Exclusion Criteria:

* 1.Patients with distant metastasis (M1) or invasion of surrounding organs
* 2.History of esophagectomy and gastrectomy (including endoscopic mucosal resection/endoscopic submucosal dissection for gastric cancer and esophageal cancer)
* 3.History of other malignant tumors within 5 years
* 4.The researcher believes that the patient is not suitable to participate in the clinical trial
* 5.Patients who persist in withdrawing from clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years after surgery
  Proportion of patients without tumor recurrence from surgery to the end of the 3-year follow-up

SECONDARY OUTCOMES:
The rate of R0-resection | About 10 days after surgery
  The proportion of patients undergoing radical resection in all surgical patients
The number of lymph node dissections and the positive | About 10 days after surgery
  The number of lymph node dissections and the positive
The duration of postoperative hospitalization | Within 6 months after surgery
  Time from end of surgery to discharge
The incidences of early postoperative complications | Within 30 days after surgery
  The incidence of postoperative complications such as pneumonia, pleural effusion, anastomotic stenosis, anastomotic leakage, duodenal stump fistula, pancreatic fistula, abdominal abscess, and deep vein thrombosis (%).
The incidence of perioperative mortality | Within 30 days after surgery
  The incidence of death due to the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Song Q, Li X, Wu D, Li S, Xie T, Lu Y, Zhang L, Xu Z, Liu L, Guo X, Wang X. The abdominal-transhiatal surgical approach versus the thoracoabdominal surgical approach in Siewert type II adenocarcinoma of the esophagogastric junction: protocol for a multicenter prospective, open, parallel, and randomized controlled trial. BMC Cancer. 2022 Mar 24;22(1):318. doi: 10.1186/s12885-022-09375-w. PMID 35331180